CLINICAL TRIAL: NCT01143155
Title: Clinical Failure and Cardiovascular Events in Hospitalized Patients With Community-Acquired Pneumonia: The Failcap Study
Brief Title: Failure and Cardiovascular Events in Community-acquired Pneumonia
Acronym: FAILCAP
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Francesco Blasi, Professor, University of Milan
Other Study IDs: FAILCAP
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; Community-acquired pneumonia; Healthcare-associated pneumonia; Failure; Cardiovascular events; Outcome
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Sputum Blood Exhaled Breath Condensate Tracheal Aspirate Pleural effusion Bronchoalveolar lavage Nasopharyngeal swabs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although failure and mortality are the most relevant outcomes in patients with Community-acquired Pneumonia (CAP), there is little discussion in the literature on their incidence and etiology. A pathophysiological approach has been recently developed and used to evaluate clinical failure in CAP patients. Clinical failure has been analyzed as related versus unrelated to CAP, considering the role that the pulmonary infection and the inflammatory response played in the development of this outcome. Cardiac events were identified as triggers of clinical failures in a significant percentage of CAP patients. The development of cardiovascular events have been also identified in CAP patients both on admission to the hospital and during hospitalization. However, data on this topic belong to studies evaluating only selected populations of veteran patients with CAP. Understanding clinical failure, as well as cardiovascular events in hospitalized patients with CAP would be useful in order to prevent complications during the hospitalization, to develop new treatment modalities and, thus, to improve outcomes.

The objectives of this international, multicenter, observational, prospective cohort study will be: 1) To define incidence, timing, etiology and risk factors of clinical failure, related vs. unrelated to CAP, in hospitalized patients with CAP; 2) To define incidence, timing, and risk factors for cardiovascular events either on hospital admission or during hospitalization in hospitalized patients with CAP.Consecutive adult patients hospitalized for CAP in acute care hospitals in Europe and US will be enrolled. Daily clinical evaluations. Demographics, history, clinical, radiological, and antibiotic therapy data will be recorded, as well as serum, urinary and respiratory samples will be collected both on admission and during hospitalization from consenting individuals. Patients will be classified as having a CAP-related versus CAP-unrelated failure, according to a pathophysiological classification. Patients will be also classified as having or not a cardiovascular event either on admission or during hospitalization.The following outcomes will be measured:

1) Incidence, timing, etiology and risk factors of clinical failure related vs. unrelated to CAP; 2) Incidence, timing and risk factors of cardiovascular events; 3)time to clinical stability, length of hospital stay, mortality at hospital discharge, and mortality at 30 and 180 days.

ELIGIBILITY:
Inclusion Criteria:

1) Signed inform consent to participate in the study

2) Criteria for community-acquired pneumonia:

1. New pulmonary infiltrate seen on chest radiograph or CT Scan of the chest within 48 hours after hospitalization.

   plus at least one of the following:
2. New or increased cough with/without sputum production
3. Fever (documented temperature -rectal or oral- > 38.3 or hypothermia (documented temperature -rectal or oral- < 36 C)
4. Evidence of systemic inflammation (such as abnormal white blood cell count -either leukocytosis (> 10,000/cm3) or leukopenia (< 4,000/cm3) - or C-reactive protein (CRP) or procalcitonin (PCT) values above the local upper limit.

3) Patients with a diagnosis of healthcare-associated pneumonia (HCAP) will be included in the study and a secondary analysis will performed on this subgroup of patients.

Exclusion Criteria:

Patients who meet at least one of the following definitions will be excluded from the analysis:

1. Patient has hospital-acquired pneumonia, defined as pneumonia that develops after 48 hours of the current hospitalization, or pneumonia that develops in a patient who had been discharged from the hospital within the prior 14 days of the current hospitalization.
2. Patient is re-admitted with a new episode of pneumonia during the 14-day follow up period from the previous hospitalization.
3. Unstable psychiatric or psychological condition rendering the subject unlikely to be cooperative or to complete the study requirements.
4. Subject history that in the investigator's opinion would preclude subject compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to any of the study centers will be screened for study entry. Patients with a diagnosis of community-acquired pneumonia (including those with health-care associated pneumonia) will be evaluated to define study entry criteria
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clinical failure | 30 days
  Incidence rates for clinical failure will be standardized and reported. Statistically significant differences between clinical failure related vs. unrelated to CAP will be investigated. Timing of clinical failure rates for those with clinical failure related vs. unrelated to pneumonia will be standardized and reported. Etiology and risk factors of clinical failure will be investigated through linear models, in order to identify associations of factors with the outcome and possible independent groups of factors in the explanation of the outcome.

SECONDARY OUTCOMES:
Cardiovascular event | 30 days
  Incidence rates for each cardiovascular event will be reported and standardized. Etiology and risk factors of cardiovascular events will be investigated through linear models.
Time to clinical stability | 7 days
  A patient will be considered to reach clinical stability when the following criteria will be met in a single day during hospitalization: 1) improved clinical signs (cough and shortness of breath); 2) patient will be afebrile for at least eight hours; 3) improving leukocytosis (decreased at least 10% from the previous day) or PCR or PCT 4) tolerating oral intake. Criteria for clinical stability will be evaluated daily during the first seven days of hospitalization.
Length of hospital stay | 30 days
  Number of days from the date of admission to the date of discharge.
In-hospital mortality | 30 days
  In-hospital mortality will be considered if death by any cause will occur during hospitalization. Patients will be followed from day of admission to day 30; those who remain hospitalized for more than 30 days will be considered alive.
Adverse events after hospital discharge | up to 180 days after hospital discharge
  Data after hospital discharge will be collected during either a visit at clinics or a phone call performed at 30 and 180 days after the diagnosis of CAP was made. Adverse events will be considered if either death, CAP-related vs. CAP-unrelated, or re-hospitalization, CAP-related vs. CAP-unrelated, will occur within 180 days after hospital discharge. In addition, data regarding visits at general practitioner clinic, antibiotic use, cardiovascular events, discharge setting (nursing home, intermediate care facility, home) will be also collected.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Blasi, M.D., PhD, Study Director — Dipartimento toraco-polmonare e cardio-circolatorio, University of Milan, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy; Stefano Aliberti, M.D., Principal Investigator — Respiratory Department, AO San Gerardo, University of Milan-Bicocca, Monza, Italy; Julio Ramirez, M.D., Study Director — Division of Infectious Diseases, Department of Medicine, University of Louisville, Louisville, Kentucky, USA; Roberto Cosentini, M.D., Principal Investigator — Emergency Medicine Department, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy; Vincenzo Valenti, M.D., Principal Investigator — UO Pneumologia, IRCCS Policlinico San Donato, University of Milan, Milan, Italy; Antonio Voza, M.D., Principal Investigator — UO Medicina d'Urgenza, Istituto Clinico Humanitas; Milan, Italy; Delfino Legnani, M.D., Principal Investigator — UO Pneumologia, Ospedale "Luigi Sacco", University of Milan, Milan, Italy; Alberto Pesci, M.D., Principal Investigator — Clinica Pneumologia, Azienda Ospedaliera S. Gerardo di Monza, University of Milano-Bicocca, Monza, Italy; Luca Richeldi, M.D., Principal Investigator — Department of Respiratory Disease, University of Modena and Reggio Emilia, Modena, Italy; Daiana Stolz, M.D., MPH, Principal Investigator — Clinic of Pneumology, University Hospital Basel, Petersgraben 4, CH-4031 Basel, Switzerland; Paula Peyrani, M.D., Principal Investigator — Division of Infectious Diseases, University of Louisville, KY; USA
Locations (1):
- Dipartimento toraco-polmonare e cardio-circolatorio, University of Milan, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Niederman MS, Mandell LA, Anzueto A, Bass JB, Broughton WA, Campbell GD, Dean N, File T, Fine MJ, Gross PA, Martinez F, Marrie TJ, Plouffe JF, Ramirez J, Sarosi GA, Torres A, Wilson R, Yu VL; American Thoracic Society. Guidelines for the management of adults with community-acquired pneumonia. Diagnosis, assessment of severity, antimicrobial therapy, and prevention. Am J Respir Crit Care Med. 2001 Jun;163(7):1730-54. doi: 10.1164/ajrccm.163.7.at1010. No abstract available. PMID 11401897
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Aliberti S, Amir A, Peyrani P, Mirsaeidi M, Allen M, Moffett BK, Myers J, Shaib F, Cirino M, Bordon J, Blasi F, Ramirez JA. Incidence, etiology, timing, and risk factors for clinical failure in hospitalized patients with community-acquired pneumonia. Chest. 2008 Nov;134(5):955-962. doi: 10.1378/chest.08-0334. Epub 2008 Jun 26. PMID 18583514
- [Background] Ramirez J, Aliberti S, Mirsaeidi M, Peyrani P, Filardo G, Amir A, Moffett B, Gordon J, Blasi F, Bordon J. Acute myocardial infarction in hospitalized patients with community-acquired pneumonia. Clin Infect Dis. 2008 Jul 15;47(2):182-7. doi: 10.1086/589246. PMID 18533841
- [Background] Musher DM, Rueda AM, Kaka AS, Mapara SM. The association between pneumococcal pneumonia and acute cardiac events. Clin Infect Dis. 2007 Jul 15;45(2):158-65. doi: 10.1086/518849. Epub 2007 Jun 6. PMID 17578773
- [Background] Jasti H, Mortensen EM, Obrosky DS, Kapoor WN, Fine MJ. Causes and risk factors for rehospitalization of patients hospitalized with community-acquired pneumonia. Clin Infect Dis. 2008 Feb 15;46(4):550-6. doi: 10.1086/526526. PMID 18194099
- [Background] Mortensen EM, Coley CM, Singer DE, Marrie TJ, Obrosky DS, Kapoor WN, Fine MJ. Causes of death for patients with community-acquired pneumonia: results from the Pneumonia Patient Outcomes Research Team cohort study. Arch Intern Med. 2002 May 13;162(9):1059-64. doi: 10.1001/archinte.162.9.1059. PMID 11996618